CLINICAL TRIAL: NCT07079839
Title: Threat-related Sensory Cortical (SC) Disinhibition and SPA Pathology in Posttraumatic Stress Disorder (PTSD) (Aim 3; Expts. 2&3)
Brief Title: A Neurosensory Account of Anxiety and Stress (Study 2)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Wen Li, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-23-1106 (study 2); R01MH132209 (NIH)
Record Dates: First submitted 2025-07-09; First posted 2025-07-23 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Threat-related Sensory Cortical (SC) Disinhibition; Posttraumatic Stress Disorder (PTSD)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Transcranial Alternating Current Stimulation (tACS) (Experimental)
  Interventions: Device: Transcranial Alternating Current Stimulation (tACS)
- Sham for Transcranial Alternating Current Stimulation (tACS) (Sham Comparator)
  Interventions: Device: Sham for Transcranial Alternating Current Stimulation (tACS)
- Active Control - Transcranial Random Noise stimulation (tRNS) (Active Comparator)
  Interventions: Device: Transcranial Random Noise stimulation (tRNS)

INTERVENTIONS:
Device: Transcranial Alternating Current Stimulation (tACS) — A weak electrical current will be passed through the scalp over targeted cortical regions via a transcranial electrical stimulation system (Soterix Medical, Inc), for a span of 10 to 40 minutes at a time. Participants will receive a 2 milliamp (mA) sinusoidal current oscillating at individual participants' baseline peak alpha frequencies (PAF; 7-13 Hz), which will be determined by a 3-min resting state EEG recording during the setup. Current intensities will be modified to address individual participants' subjective reports of discomfort, with a maximum intensity of 2 mA. Stimulation electrodes will be placed within an EEG cap fitted over the participant's head.
  Arms: Transcranial Alternating Current Stimulation (tACS)
Device: Sham for Transcranial Alternating Current Stimulation (tACS) — Stimulation electrodes will be placed on the scalp, but no current will be passed. Stimulation electrodes will be placed within an EEG cap fitted over the participant's head.
  Arms: Sham for Transcranial Alternating Current Stimulation (tACS)
Device: Transcranial Random Noise stimulation (tRNS) — A weak electrical currents will be passed through the scalp over targeted cortical regions via a transcranial electrical stimulation system (Soterix Medical, Inc), for a span of 10 to 40 minutes at a time. Participants will receive a 2 mA sinusoidal current oscillating at random frequency (1-200 Hz). Current intensities will be modified to address individual participants' subjective reports of discomfort, with a maximum intensity of 2 mA. Stimulation electrodes will be placed within an EEG cap fitted over the participant's head.
  Arms: Active Control - Transcranial Random Noise stimulation (tRNS)

SUMMARY:
This study will take a basic neuroscience approach to investigate pathological mechanisms underlying PTSD. Additionally, the study aims to identify how Transcranial Alternating Current Stimulation (tACS) brain stimulation can modulate and correct neural networks and related emotions of anxious arousal and hypervigilance, with the goal of assessing tACS brain stimulation technology as a novel intervention for symptoms of anxiety.

DETAILED DESCRIPTION:
This study includes experiments 2 & 3 to address Aim 3--threat-related SC disinhibition and Sensory-Prefrontal-cortex-Amygdala (SPA) pathology in PTSD. The goal of this study is to develop and test a novel pathophysiology of PTSD by integrating sensory cortical (SC) and amygdala-prefrontal cortex (PFC) dysfunctions into a tripartite Sensory-Prefrontal-Cortex-Amygdala (SPA) model. The investigators will recruit 80 healthy subjects and 80 patients with PTSD in a randomized, double-blind, controlled design, where they be randomly assigned to 1) Transcranial Alternating Current Stimulation (tACS) at individual alpha peak frequency (active condition); 2) sham control tACS; or 3) active control, which will be transcranial random noise stimulation (tRNS) (random frequency 1-200 Hz). Simultaneous EEG/fMRI recordings and behavioral responses will be acquired before and after tACS/sham tACS/tRNS stimulation. During tACS/sham tACS/tRNS stimulation, stimulation electrodes will be placed inside the holders of an EEG cap attached to the head of the participant. Experiments 2 & 3 include a visual search task and an olfactory detection task, respectively, and both experiments include threat and neutral stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* With normal or corrected-to-normal vision and normal olfaction
* Between the ages of 18 and 50 years
* Meeting the tACS screening criteria (see List I below; e.g., lack of a serious head injury or loss of consciousness)
* Patients: Diagnosis of PTSD
* Patients: If taking psychotropic medications, medication stability in the past 2 months
* If having mild substance use disorder (for patients) or occasional substance use, abstention from use 48 hours before the experiment.

Exclusion Criteria:

* A history of diagnosis for a major medical illness (e.g., cancer, metabolic syndrome, cardiovascular disease, inflammatory disorders) or a neurological disorder (e.g., seizure, stroke, Parkinson's disease).
* Patients: Concurrent Axis I diagnosis (depression, anxiety, and mild substance use disorder are allowed given their high comorbidity with PTSD).
* Healthy controls: A history of diagnosis for a Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 Axis I disorder or current use of psychoactive medications.
* Severe psychiatric instability or severe situational life crises, including evidence of being actively suicidal or homicidal, or any behavior that poses an immediate danger to self or others.
* History of head trauma with unconsciousness (> 5 minutes)
* Report that they regularly drink 3 or more alcoholic beverages a day.
* Report that they are unable to abstain from substance use (including alcohol, nicotine, cannabis, amphetamines, narcotics, solvents, cocaine, hallucinogens, tranquilizers, barbiturates, etc.) or sleep medication for 48 hours before being scanned.
* Are on calcium channel blockers (e.g., verapamil, nifedipine) or alpha-blockers (e.g., prazosin, terazosin) and are unable to stop these medications for a 48-hour period prior to scanning (to exclude the impact of these medications on the interpretation of fMRI/EEG).
* Failed Urine Drug Screening Test: A rapid urine screening test that utilizes monoclonal antibodies to detect elevated levels of specific drugs (including alcohol, amphetamines, benzodiazepines, barbiturates, cocaine, marijuana, opiates, etc.) in urine (iCup)
* Pregnancy based on urine test. The safety of magnetic resonance (MR) systems has not been established for fetuses
* Having electrically, magnetically, or mechanically activated implants (e.g., cardiac pacemakers), because the electromagnetic fields produced by the MR system may interfere with the operation of these devices.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in neural oscillatory activity as assessed by electroencephalogram (EEG) alpha power change | baseline (pre-stimulation); immediately post-stimulation (about 10 to 40 minutes after start of stimulation)
Change in cortical activity as assessed by functional magnetic resonance imaging (fMRI) blood-oxygen-level-dependent (BOLD) signal change | baseline (pre-stimulation); immediately post-stimulation (about 10 to 40 minutes after start of stimulation)

SECONDARY OUTCOMES:
Change in visual search as assessed by change in percent accuracy on the visual search experiment | baseline (pre-stimulation); immediately post-stimulation (about 10 to 40 minutes after start of stimulation)
Change in visual search as assessed by change in reaction time on the visual search experiment | baseline (pre-stimulation); immediately post-stimulation (about 10 to 40 minutes after start of stimulation)
Change in olfactory detection as assessed by change in percent accuracy on the olfactory detection experiment | baseline (pre-stimulation); immediately post-stimulation (about 10 to 40 minutes after start of stimulation)
Change in olfactory detection as assessed by change in reaction time on the olfactory detection experiment | baseline (pre-stimulation); immediately post-stimulation (about 10 to 40 minutes after start of stimulation)
Change in salience detection and vigilance behavior as assessed by skin conductance measured in microsiemens (μS) | baseline (pre-stimulation); immediately post-stimulation (about 10 to 40 minutes after start of stimulation)

CONTACTS AND LOCATIONS:
Overall Officials: Wen Li, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Starting 6 months after publication.
Access Criteria: All researchers.